CLINICAL TRIAL: NCT01664780
Title: Acoustic Radiation Force Impulse Imaging (ARFI) in Patients After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: ARFI-UK Erlangen
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Liver Transplantation
Keywords: standard; values; share; wave velocity; in ARFI imaging
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients after liver transplantation
  Interventions: Device: ARFI imaging

INTERVENTIONS:
Device: ARFI imaging

SUMMARY:
Aims: Prospective evaluation of the applicability of acoustic radiation force impulse(ARFI) imaging to assess liver fibrosis in patients after orthotopic liver transplantation.

Material and methods: We prospectively assess the performance of ARFI imaging in planned 100 patients after orthotopic liver transplantation. We evaluate shear wave velocity of the left and right liver lobe with the convex array (6C1HD)ultrasound transducer and compare the results with clinical data and B-mode criteria.

ARFI elastometry is an increasingly popular non-invasive method for the assessment of hepatic fibrosis and cirrhosis. To date, ARFI technology has not been applied systematically in patients after orthotopic liver transplantation. Therefore we want to establish standard values in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients after orthotopic liver transplantation.

Exclusion Criteria:

* Patients without status after orthotopic liver transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after orthotopic liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dane Wildner, MD, Principal Investigator — Dep. of Medicine 1, University of Erlangen-Nuremberg
Locations (1):
- University Hospital of Erlangen, Dep. of Medicine 1, Erlangen, Germany